CLINICAL TRIAL: NCT06673186
Title: Patient Satisfaction and Prosthetic Complications of Bar Locator Versus Bar Clip Attachments for Mandibular Two-Implant Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Wageh Abozaed Elsaed Mansour, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: M21011122
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Edentulism
MeSH Terms: interventions — Denture, Overlay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (bar locator): Patients were given overdentures with bar locator attachments (Experimental): Group I received mandibular overdentures with a bar locator attachment , specially designed milled bar with parallel walls was built for this group, and two holes were drilled in the top surface of the bar using a 1.7 mm bar drill to create the threaded site in the waxed bar, followed by a 2.0 mm bar tap. The locator female component was then connected to the corresponding site using a customised rider.
  Interventions: Other: overdenture
- group2, Patients were given overdentures with bar clip attachment. (Experimental): bar clip attachment. Patients received mandibular overdentures with bar clip attachments. A plastic prefabricated bar was cast in cobalt-chrome alloy. Group II patients received mandibular overdentures with bar clip attachments. A plastic prefabricated bar was cast in cobalt-chrome alloy.
  Interventions: Other: overdenture

INTERVENTIONS:
Other: overdenture — Patient satisfaction (primary outcome) was measured by a visual analog scale (VAS). OHRQoL (secondary outcome) was measured by oral health impact profile (OHIP-14). Questions of VAS and OHIP-14 were evaluated after 3 months The patients were divided into two equal groups.

SUMMARY:
Purpose: This study evaluated patient satisfaction and oral health-related- quality of life (OHRQoL) with implant overdentures retained with bar locator versus bar clip attachment for mandibular two-implant overdentures. Materials and methods: This study included sixteen edentulous patients. Every patient received new maxillary and mandibular dentures. Two dental implants have been embedded in the mandibular canine areas. The participants were randomly divided into two equal groups: Group I (bar locator): Patients were given overdentures with bar locator attachments, Group II (bar clip): Patients were given overdentures with bar clip attachment. Patient satisfaction (primary outcome) was measured by a visual analog scale (VAS). OHRQoL (secondary outcome) was measured by oral health impact profile (OHIP-14). Questions of VAS and OHIP-14 were evaluated after 3 months.

The aim of this study was to document and report on the prosthetic complications associated with mandibular implant overdentures using bar locator and bar clip attachments. The study aimed to test the null hypothesis that the complications would not differ based on the type of retention (locator or clip).

ELIGIBILITY:
Inclusion Criteria:

* Each patient had sufficient remaining alveolar ridge in the upper and lower jaw to support implants in the lower jaw area
* a minimum length of 11 mm and a diameter of 3.7 mm, as confirmed by cone beam computed tomography.
* patient had a class I jaw relationship
* adequate space between the arches.
* healthy, firm gum tissue.

Exclusion Criteria:

* participants with uncontrolled diabetes,
* heavy smoking
* drinking habits
* temporomandibular joint (TMJ) issues.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Patient satisfaction (primary outcome) was measured by a visual analog scale (VAS). OHRQoL (secondary outcome) was measured by oral health impact profile (OHIP-14). Questions of VAS and OHIP-14 were evaluated after 3 months.
  Patient Satisfaction
prosthetic complications | Mechanical complications were clinically examined and included Distortion /wear of retentive components, Bar screw loosening, Fracture of opposing prosthesis, Teeth wear, Fracture at the midline of the prosthesis and Teeth separation within 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Wageh Abozaed, Al Mansurah, Egypt